CLINICAL TRIAL: NCT05372770
Title: Pilot Study to Observe Effects of Using Flourish Vaginal Care System to Establish Neovaginal Microbiome After Gender-Confirmation Surgery
Brief Title: Flourish Vaginal Care System to Establish Neovaginal Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vaginal Biome Science (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NV0122
Record Dates: First submitted 2022-05-09; First posted 2022-05-13 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Neovaginal Microbiome
Keywords: neovagina; microbiome; lactobacillus; transgender; probiotic

STUDY DESIGN:
Intervention Model Description: Two groups of transgender women who have undergone surgery plus a group of healthy cisgender women who have not undergone surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Group 1: Transgender women using Flourish (Experimental): After gender-confirming surgery, this group will use the Flourish Vaginal Care System for six months, ramping up usage with healing. They will use "Balance" external wash beginning day 6 after surgery; "Restore®" vaginal moisturizing gel on dilators beginning day 6 after surgery; Restore every other day at bedtime with "BiopHresh" homeopathic/probiotic suppository every 3rd day at bedtime beginning week 6 after surgery through end of study at 6 months.
  Interventions: Device: Flourish Vaginal Care system
- Group 2: Transgender women not using Flourish (No Intervention): After gender-confirming surgery, this group will use only KY jelly on dilators beginning day 6 after surgery according to routine care; they will use any standard hygiene product (soap, body wash, etc) of their choice except products used by Group 1 through the end of the study at 6 months.
- Group 3: Cisgender women (Other): This group will use the Flourish Vaginal Care system for 6 months: Balance external wash daily; Restore intravaginal gel every other day at bedtime; BiopHresh homeopathic/probiotic suppository every 3rd day at bedtime through the end of study.
  Interventions: Device: Flourish Vaginal Care system

INTERVENTIONS:
Device: Flourish Vaginal Care system — Flourish includes Restore® vaginal moisturizing gel, a Class II medical device cleared by the FDA, in addition to two other kit components
  Arms: Group 1: Transgender women using Flourish; Group 3: Cisgender women

SUMMARY:
This study examines whether use of a commercially-available vaginal wellness system is able to establish a microbiome in transgender women.

DETAILED DESCRIPTION:
Very little is known about the neovaginal microbiome, but it has been described as being a polymicrobial state similar to bacterial vaginosis (BV) in cis women. The Flourish Vaginal Care System is a commercially-available over-the-counter vaginal wellness kit that helps relieve symptoms of BV. This study is intended to determine whether that kit could also help transgender women who have recently undergone gender-confirming surgery to establish a neovaginal microbiome that is dominated by lactobacilli, as observed in healthy cis women. This could increase health and subjective satisfaction of the neovagina. This study examines the (neo)vaginal microbiome in transgender women with and without using Flourish, as well as a group of healthy cisgender women.

ELIGIBILITY:
Inclusion Criteria:

1. Transgender women over age 18 who are preparing to undergo gender-confirmation surgery.
2. Healthy cisgender women ages 18-52

Exclusion Criteria:

1. Immunosuppressed
2. Known allergies or sensitivities to aloe vera or to other components of Restore®, Balance, or BiopHresh®
3. Known (neo)vaginal infection that is not yeast or BV at start of protocol
4. Inability to tolerate Restore gel by day 13 after surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Individuals must be either 1) transgender women who are undergoing gender-confirming surgery; or 2) cisgender women
Enrollment: 56 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Vaginal microbiome | Collections at time 0, 6 weeks, and 6 months
  Observation of changes in the composition of the vaginal fluid microbiome over six months using commercially available next-generation sequencing kit (16s rRNA). Biomes will be categorized to "community state type" (Ravel 2011), and genus- or species-level relative abundance will be compared.
Vaginal pH | Collections at time 0, 6 weeks, and 6 months
  Observation of changes in vaginal pH over six months by pH strip

SECONDARY OUTCOMES:
VSQ | Collections at time 0, 6 weeks, and 6 months
  Responses to the Vulvovaginal Symptoms Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Christine McGinn, DO, Principal Investigator — Papillon Center
Locations (1):
- Papillon Wellness Center, New Hope, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No